CLINICAL TRIAL: NCT00488020
Title: the Use of Autogenous Adult Stem Cells in the Treatment of Critical Ischemia
Brief Title: Stem Cells for Treating Critical Ischemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto de Molestias Cardiovasculares (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: imc1
Record Dates: First submitted 2007-06-15; First posted 2007-06-19 (Estimated); Last update posted 2008-06-13 (Estimated); Status verified 2007-06

CONDITIONS: Critical Limb Ischemia; Ischemic Ulcers
Keywords: rest pain; ischemic ulcers
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: stem cells transplant

SUMMARY:
Collection of bone marrow blood Selection of mononuclear cells dilution with albumin injection into the calf muscles through 40 shots

DETAILED DESCRIPTION:
About 500cc of blood are collected from the iliac bone marrow under epidural anesthesia.In the cell therapy lab this blood is harvested and mononuclear cells are separated.This procedure takes roughly 4 hours.After dilution in albumin (40cc)the mononuclear cells are injected into the calf muscles through 40 shots.This procedure is indicated for patients with lower limb ischemia on whom all the others known therapies have failed

ELIGIBILITY:
Inclusion Criteria:

* Fontaine's classification grade 3 and 4 patients

Exclusion Criteria:

* Record of cancer in the last 5 years
* Over 80 years
* Diabetic retinopathy

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2006-04; Study Completion 2007-06 (Estimated)

PRIMARY OUTCOMES:
Suppress pain and heal ischemic ulcers | 6 months

SECONDARY OUTCOMES:
improve quality of life | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jose D Araújo, MD, Principal Investigator — Instituto de Molestias Cardiovasculares
Locations (1):
- Instituto de Molestias Cardiovasculares, São José do Rio Preto, São Paulo, Brazil